CLINICAL TRIAL: NCT00355823
Title: Phase I Study of the Electric Field Near Human Skin Wounds
Brief Title: Bioelectric Field Imaging Near Human Skin Wounds
Status: Completed | Type: Observational
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Antoinette F. Hood, Eastern Virginia Medical School
Other Study IDs: BFI and wounds; R44GM069194-03 (NIH)
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2006-11

CONDITIONS: Wounds
Keywords: electric field; wound current; wound healing; bioelectric field; chronic ulcer; diabetic; Diabetes; aging
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators have developed a new non-invasive medical device called the Bioelectric Field Imager. They plan to use this device to measure the electric field near small lancet wounds in 60 volunteers. Their hypothesis is that the electric field is an early stimulus for wound healing and the magnitude of this field will vary with wound healing capability. The investigators will compare the electric fields near arm and leg wounds in males and females in the age groups of 18-30 and 65-80. In addition they will measure these wound fields in diabetics and near chronic ulcers.

DETAILED DESCRIPTION:
We will first characterize the lateral electric field near reproducible skin wounds in healthy male and female subjects 18-30 years of age. A standard superficial, dermal wound 0.5 mm long will be inflicted using the Ascensia Microlet Vaculance by Bayer Health Care with a 21 gauge lancet on its deepest setting. This setting will penetrate the epidermis and stop within the dermis. We will first determine variability within the same individual by measuring the electric field near two wounds close to each other on the volar forearm. We will then determine the variability between different body regions by comparing the wound field near a lancet wound in the volar forearm and one in the leg. If hair is present it will be removed by shaving the wound site prior to wounding. By collecting these data from 10 males and 10 females in both age groups we can determine if there is a gender or age dependence to the field strength. Finally we will determine the lateral electric field near lancet wounds in diabetics and near chronic skin wounds. If these fields are smaller than fields found near acute wounds, it would provide a rationale for future studies imposing electric fields to enhance wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years or 65-80 years
* Chronic leg ulcer present
* Diabetic

Exclusion Criteria:

* Hemophilia
* Fever

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two age groups will be studied: 1. Young adults 18-19 years old; and 2. older adults 65-80 years old.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette F. Hood, M.D., Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Virginia Clinical Research, Inc., Norfolk, Virginia, United States